CLINICAL TRIAL: NCT04800198
Title: Intraoral Measurement of Pressure in Preterm Infants
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Helmut Küster, MD, Principal Investigator, University Medical Center Goettingen
Other Study IDs: 1
Record Dates: First submitted 2021-03-03; First posted 2021-03-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Preterm Infants
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: non-invasive ventilation — none, measurements only

SUMMARY:
The aim of the study is to show pressure curves in the nasopharynx in non-invasively ventilated and spontaneously breathing premature and newborn babies

DETAILED DESCRIPTION:
The aim of the investigation is to show the pressure curves in the nasopharynx in non-invasively ventilated and spontaneously breathing premature and newborn babies, with a number large enough for an analysis. For this purpose, the pressure in the nasopharynx of these children is to be measured using a suction catheter, as is usually used to suction off mucus and saliva, and the measured values are to be evaluated with software. This method is a tried and tested method in adults for measuring the pressure conditions in the nasopharynx, which was developed and used by Mr. Olthoff. A possible later clinical application in premature and newborn infants ranges from the measurement of breathing and ventilation to manual control of respiratory support depending on the measured value to automatic triggering and control of a ventilator in the sense of nSIPPV ventilation (non-invasive synchronized intermittent positive pressure ventilation )

ELIGIBILITY:
Inclusion Criteria:

newborns, non-invasive ventilation

Exclusion Criteria:

* Bad clinical condition of the patient (e.g. sepsis)
* Bleeding tendency
* Anatomical peculiarities that make it difficult to insert the suction catheter through the nose (e.g. choanal atresia)
* Lack of acceptance of the probe by the child
* Proven infection / colonization of the child by a multi-resistant germ (MRGN 2-4, MRSA) or with noro- / adenoviruses
* Missing / withdrawn consent by the legal guardians

Ages: 3 Days to 3 Months | Sex: All
Age Groups: Child
Study Population: newborns, in hospital
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Median Pressure reached by any tape of non-invasive ventilation | 1 year
  The pressure reached by non-invasive ventiation (nCPAP or HFT) in neonates of any gestation is measured weekly to collect data on how to correctly set the ventilator.

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Küster, MD, Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medicine Göttingen, Göttingen, Germany